CLINICAL TRIAL: NCT01486680
Title: Prospective Randomised Controlled Trial Comparing the Efficacy of Laparoscopic Silastic Ring Roux-en-Y Gastric Bypass Versus Laparoscopic Sleeve Gastrectomy for the Management of Type 2 Diabetes Mellitus in Obese Patients
Brief Title: Silastic Ring Gastric Bypass Versus Sleeve Gastrectomy for Type 2 Diabetes Mellitus in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Shore Hospital, New Zealand (Other)
Responsible Party: Principal Investigator, Dr. Michael Booth, Consultant Bariatric, Upper GI and General Surgeon, North Shore Hospital, New Zealand
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NTY/11/07/082; ACTRN12611000751976 (Registry Identifier: Australian New Zealand Clinical Trials Registry)
Record Dates: First submitted 2011-11-28; First posted 2011-12-06 (Estimated); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Type 2 Diabetes Mellitus; Obesity
Keywords: Gastric bypass; Silastic ring gastric bypass; Roux-en-Y gastric bypass; Sleeve gastrectomy; Body composition analysis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laparoscopic Silastic Ring Roux-en-Y Gastric Bypass (Active Comparator)
  Interventions: Procedure: Laparoscopic Silastic Ring Roux-en-Y Gastric Bypass
- Laparoscopic Sleeve Gastrectomy (Active Comparator)
  Interventions: Procedure: Laparoscopic Sleeve gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic Silastic Ring Roux-en-Y Gastric Bypass — An isolated lesser curve-based gastric pouch will be created, with an antecolic antegastric Roux limb fashioned measuring 100 cm in length. The biliopancreatic limb will measure 50cm for all patients. A 6.5cm silastic ring will be placed above the gastrojejunostomy to prevent long term stomal dilatation.
  Other Names: Silastic ring Gastric bypass; Fobi pouch; RYGB; LRYGBP; LRYGB; GBP; SR gastric bypass
  Arms: Laparoscopic Silastic Ring Roux-en-Y Gastric Bypass
Procedure: Laparoscopic Sleeve gastrectomy — Resection of the greater curvature of the stomach from the distal antrum (2cm proximal to pylorus) to the angle of His, using a laparoscopic stapling device over a 36Fr bougie, will be performed to create a lesser curve gastric sleeve
  Other Names: Vertical sleeve gastrectomy
  Arms: Laparoscopic Sleeve Gastrectomy

SUMMARY:
Type 2 diabetes (T2DM) and obesity are becoming increasingly common in New Zealand (NZ) and worldwide. Both are associated with a risk of early mortality (death). Whilst weight loss surgery is known to be effective for weight loss, current research suggests that it may also be effective in resolving T2DM in around 60-80% of patients, with some no longer requiring their medication. The mechanism for this remains unclear.

Two main types of weight loss surgery are performed in NZ public hospitals, which include gastric bypass and sleeve gastrectomy. The gastric bypass is a more complex procedure compared to the sleeve gastrectomy. Whilst both appear to be effective for weight loss (with most patients losing more than 60% of their excess weight), it is still not known which one is better for treating T2DM.

This study will therefore compare which of these two surgical procedures is most effective at treating T2DM in obese patients, as well as comparing whether there are any differences in the amount of weight lost, side effects and quality of life.

DETAILED DESCRIPTION:
EFFECTS OF DIABETES AND OBESITY The World Health Organization indicates that 346 million people worldwide have diabetes. This is expected to double between 2005 and 2030. Type 2 diabetes mellitus (T2DM) accounts for 90% of people with diabetes and is known to result from a combination of physical inactivity and excess weight. In New Zealand (NZ) more than 200,000 people have diabetes, with an incidence amongst the Maori and Pacific population three times greater than other NZ ethnic groups. Obesity is also more prevalent amongst this population, with each 5 kg/m2 higher BMI resulting in a 30% higher overall mortality.

Over the last 10 years bariatric surgery has been recognised as an effective strategy to treat both morbid obesity and T2DM. Indeed in a systematic review in 2004, by Buchwald et al, an overall T2DM remission rate of 76% was seen following bariatric surgery. In March 2011 the International Diabetic Federation released a position statement recognising bariatric surgery as an appropriate treatment option in those patients with T2DM and a body mass index (BMI)> OR = 35kg/m2 or BMI 30-35kg/m2 where medical treatment has failed.

SURGICAL PROCEDURES Laparoscopic Roux-en-Y gastric bypass (LRYGB): Currently the most commonly performed bariatric procedure worldwide. It combines a restrictive and malabsorptive (duodenal bypass) component, with a mean excess weight loss (EWL) of 61.6% and T2DM remission rate of 83.8% reported. Analysis of our own series identified a T2DM remission rate at 1 year of 88%.

Laparoscopic sleeve gastrectomy (LSG): A predominantly restrictive procedure (no bypass component), which was initially used as a staged approach to biliopancreatic diversion and duodenal switch (BPD-DS), has gained increasing popularity due its relatively lower technical complexity. In a recent systematic review a mean EWL of >45% (range 6.3 - 74.6%) was reported with an overall T2DM remission rate of 66%, which reduced to 59% where only those studies reporting 1 year outcomes were analysed. There is however a lack of medium and long term data and meta-analysis is currently not feasible in view of the high heterogeneity of studies and the lack of randomised controlled trials.

MECHANISM OF ACTION The mechanism of T2DM remission following these procedures remains unclear and may relate to the effects of reduced caloric intake or gut hormone effects in the proximal and distal intestine. Following LRYGB, the improvement in glycaemic control appears to occur before weight loss and may be explained by exclusion of the duodenum / proximal jejunum reducing insulin resistance or an enhanced hormonal response resulting from nutrients in the distal small bowel. Following LSG both hormonal changes and a hindgut theory have been proposed. In addition there is increasing evidence that changes in bone mineral density and body composition, with a reduction in body fat and lean tissue mass, and an increase in resting energy expenditure, may also occur following gastric bypass and other restrictive surgical procedures. It is unclear whether such changes correlate with the degree of comorbidity resolution after surgery.

CONCLUSION At the current time much of the data relating to LSG is based on non-randomised observational studies and it remains unclear whether the promising T2DM remission rates and excess weight loss reported will be sustainable in the long term. In the only published randomised trial, by Lee et al. from Taiwan, to compare T2DM remission rates at 1 year between LSG and gastric bypass in BMI < 35, a much higher remission rate of 93% was seen following gastric bypass compared with 47% following LSG. Given the potential technical benefits of LSG, there is an urgent need to compare the efficacy of this procedure with the more commonly performed LRYGB procedure, at a time when clinical equipoise remains, in order to determine the optimum approach to T2DM in the future.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 to 50 years old
* Body mass index 35-65
* Type 2 diabetes mellitus for at least 6 months
* Suitable for either of the two surgical procedures

Exclusion Criteria:

* Aged >50 years
* BMI >65
* Type 1 diabetes mellitus or secondary forms of diabetes
* Previous bariatric or oesophagogastric surgery
* Previous small bowel resection
* Severe cardiorespiratory or gastrointestinal disease
* Myocardial infarction or cerebrovascular event within last 6 months
* Malignancy in last 5 years
* Poorly controlled psychiatric disorder
* Contraindication to general anaesthesia
* Current smoker

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2011-09; Primary Completion 2014-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Remission of type 2 diabetes mellitus/ glycaemic control | 5 years
  COMPLETE:Defined as fasting plasma glucose less than 5.6mmol/L and glycated haemoglobin (HbA1c) less than 6.0% in the abscence of active pharmacologic therapy PARTIAL:Defined as fasting plasma glucose between 5.6 and 6.9mmol/L and glycated haemoglobin (HbA1c) between 6.0 and 6.5% in the abscence of active pharmacologic therapy

SECONDARY OUTCOMES:
Comorbidity resolution | 5 years
  Measurement of changes in blood pressure, blood lipid profile, obstructive sleep apnoea symptoms and CPAP usage, urinary incontinence frequency, angina severity, reflux symptoms using Visick scale, medication changes
Peri/ post-operative morbidity and mortality | 30-day, In-hospital, 1 year and 5 years
  For example haemorrhage, thromboembolic events, cardiorespiratory events, marginal ulceration, anastomotic / staple line leak, internal herniation, nutritional deficiencies and mortality
Changes in body composition, resting energy expenditure and bone density | 1 year and 5 years
  Includes use of dual energy x-ray absorptiometry (DEXA)
Quality of Life | 1 year and 5 years
  Qualitative scores using Short Form-36 and Hospital and Anxiety depression scale

OTHER OUTCOMES:
Weight loss (excess weight loss and actual weight loss) | 5 years
  Weight loss in kiloigrams, Body mass Index change and percentage excess weight loss

CONTACTS AND LOCATIONS:
Overall Officials: Michael Booth, MBA FRACS, Principal Investigator — North Shore Hospital, Auckland, NEW ZEALAND
Locations (2):
- New Zealand (2):
  - North Shore Hospital, Auckland
  - University of Auckland, Auckland

REFERENCES:
- [Derived] Pullman JS, Plank LD, Nisbet S, Murphy R, Booth MWC. Seven-Year Results of a Randomized Trial Comparing Banded Roux-en-Y Gastric Bypass to Sleeve Gastrectomy for Type 2 Diabetes and Weight Loss. Obes Surg. 2023 Jul;33(7):1989-1996. doi: 10.1007/s11695-023-06635-x. Epub 2023 May 27. PMID 37243915
- [Derived] Kaur R, Kim D, Cutfield R, Booth M, Plank L, Murphy R. Good Glycemic Outcomes Following Bariatric Surgery Among Patients With Type 2 Diabetes, Obesity, and Low-Titer GAD Antibodies. Diabetes Care. 2021 Feb;44(2):607-609. doi: 10.2337/dc20-0804. Epub 2020 Dec 11. PMID 33310883
- [Derived] Murphy R, Clarke MG, Evennett NJ, John Robinson S, Lee Humphreys M, Hammodat H, Jones B, Kim DD, Cutfield R, Johnson MH, Plank LD, Booth MWC. Laparoscopic Sleeve Gastrectomy Versus Banded Roux-en-Y Gastric Bypass for Diabetes and Obesity: a Prospective Randomised Double-Blind Trial. Obes Surg. 2018 Feb;28(2):293-302. doi: 10.1007/s11695-017-2872-6. PMID 28840525
- [Derived] Murphy R, Evennett NJ, Clarke MG, Robinson SJ, Humphreys L, Jones B, Kim DD, Cutfield R, Plank LD, Hammodat H, Booth MW. Sleeve gastrectomy versus Roux-en-Y gastric bypass for type 2 diabetes and morbid obesity: double-blind randomised clinical trial protocol. BMJ Open. 2016 Jul 4;6(7):e011416. doi: 10.1136/bmjopen-2016-011416. PMID 27377635